CLINICAL TRIAL: NCT02622737
Title: Comparison of the Effects of Exercise by Functional Training, Stationary Bicycle and Exergame in Parkinson Disease
Brief Title: Study of the Effects of Three Exercise Programs in Parkinson's Disease
Acronym: STEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment site changed their admission policy to only more severely affected patients.
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Jamary Oliveira-Filho, Associate Professor, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE # 41228415.5.0000.5662
Record Dates: First submitted 2015-11-26; First posted 2015-12-04 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Accidental Falls; Exercise therapy; Virtual Reality Exposure Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Functional Training (Experimental): Functional exercise training program
  Interventions: Other: Functional training
- Stationary Bike (Experimental): Stationary bike training program
  Interventions: Device: Stationary bike
- Exergaming (Experimental): Virtual Reality Exposure Therapy
  Interventions: Device: Exergaming

INTERVENTIONS:
Other: Functional training — Three times per week, with 50 minutes per session, during 8 weeks of training activities involving 10 minutes of muscle stretching, 5 minutes of warm-up exercise, 30 minutes of a functional training and 5 minutes of respiratory exercises.
  Arms: Functional Training
Device: Stationary bike — Three times per week, with 50 minutes per session, during 8 weeks of training activities involving 10 minutes of muscle stretching, 5 minutes of warm-up exercise, 30 minutes of a Stationary Bike exercise and 5 minutes of respiratory exercises.
  Arms: Stationary Bike
Device: Exergaming — Three times per week, with 50 minutes per session, during 8 weeks of training activities involving 10 minutes of muscle stretching, 5 minutes of warm-up exercise, 30 minutes of a Virtual Reality exercise (performed by Xbox360 with KinectTM sensor) and 5 minutes of respiratory exercises.
  Other Names: Virtual Reality Exposure Therapy
  Arms: Exergaming

SUMMARY:
Introduction: Population aging is associated with increased prevalence of chronic diseases. Parkinson's disease (PD) is the second most common neurodegenerative disease in the world population, affecting motor function and functional independence progressively. The physiological aging promotes the gradual reduction of body weight, lung function, peripheral muscle strength, cardiopulmonary endurance and physical capacity, which increase the debilitating effects. Aging, when associated with PD, can induce loss of functionality, postural changes, further affecting the nutritional status, worsening the quality of life and functional independence of the individual. Although physical therapy is commonly applied with a variety of methodologies to PD patients, evidence for the effectiveness of these interventions is lacking.

Objective: The primary objective of the study is to compare the effects of Functional Training, Stationary Bike and Exergaming Exercises on proportion of fallers in elderly participants with PD. In addition, the secondary objectives are to compare the effects on cardiopulmonary endurance, posture, postural control, executive function, quality of life and functionality of individuals with PD.

Methodology: This is an interventional, randomized, blinded, longitudinal and prospective study. This research will be conducted in the State Reference Center for Health Care of the Elderly (CREASI). The sample will consist of 63 individuals with PD per group. The Experimental Group 1 will be submitted to Functional Training, the Experimental Group 2 with undergo training with Stationary Bike and the Experimental Group 3 will be submitted to exergame training using Xbox360 with KinectTM sensor. All the interventions will be performed three times per week, with 50 minutes per session, during 8 weeks.

DETAILED DESCRIPTION:
The original study goal was to recruit 210 subjects based on the assumption of a fall risk of 70% in the Bicycle group and 40% in either Exergaming or Functional Training groups, with 80% power and alpha=0.05.

GROUPS:

G1-Functional Training

The intensity was increased by progressive resistance with dumbbells, ankle weights, elastic bands and manual resistance.

1. Gait with obstacles: To perform this exercise hula hoops, rubber cones, plastic sticks, wood steps and mattresses were used.
2. Up and down stairs and ramp: The participant went up and down 3 steps and 1 ramp until completing 3 minutes.
3. Sitting and standing exercises: To increase the difficulty level were used manual resistance, dumbbell and unstable bases (swiss ball).
4. Side gear and shin guards: The participant performed side gait according to the physical therapist's commands.
5. Balance exercise: The participant performed balance exercises in proprioceptive platforms: balance discs, jumping beds proprioceptive tables.
6. Activities with ball: Kicking balls of different sizes and weights, alternating each foot.
7. Step exercises: Going up and down steps with the right or left foot according to cognitive commands of the physical therapist.
8. Foot tip exercises: The participant performed the exercise on flat and sloped surface with one or two feet maintaining sural triceps contraction for 5 seconds.
9. Graded reaching exercises: The exercise was performed standing and sitting. Dual task activities were performed.
10. Gait training: The participant walked around the gym following verbal commands to stop and change direction. Gait reeducation consisted of working scapular and pelvic girdle dissociation.

G2-Bicycle

Aerobic training on a stationary bicycle: The training intensity was 50% of maximum heart rate (adjusted for age - Karvonen formula) in the first week, increasing gradually to 75% in the eighth week.

First week: 50% of maximum heart rate. Second and Third weeks: 55% of maximum heart rate. Fourth and Fifth weeks: 65% of maximum heart rate. Sixth and Seventh weeks: 70% of maximum heart rate. Eighth week: 75% of maximum heart rate. The intensity was increased progressively by bike endurance (resistance) and speed.

G3-Exergaming

Physical components involved in Exergames (Virtual Reality Exposure Therapy): strength and muscular endurance, cardiorespiratory fitness, postural balance, executive function and emotional demands.

The participants did not use weights to perform the exercises in the Exergame Group. A physical therapist guided the participants to explore the correct posture and the articular range of motion using both tactile and assistive stimulus and/or verbal command during the games. Each mini-game lasts about 3-minutes, and to complete 30-minutes training, the same one or two mini-games were repeated in different levels of intensity and speed in each session. Mini-games of Kinect Advenctures! game:

* River Rush: One or two players must control the raft using their body, moving from side to side, and jumping in front of the Kinect sensor. Players must work as a team to earn as many points as possible.
* Reflex Ridge: One or two players can move freely on platforms (rollercoaster-like tracks), allowing them to dodge left and right, duck and jump over hazards as they spring forward. Jumping in place makes the platform move faster along its rail.
* 20,000 Leaks: The characters are positioned in a rectangular glass tank underwater, and each of the tank's four walls can crack and begin to leak water at any time. One or two players stand in front of the Kinect sensor and use their arms and legs - or any other body parts - to stop leaking water.

ELIGIBILITY:
Inclusion Criteria:

* Regular use of medication for PD;
* Age greater than or equal to 60 years;
* Stage 2, 2.5 or 3 according to the modified Hoehn and Yahr classification;
* Signed informed consent.

Exclusion Criteria:

* neurodegenerative diseases other than Parkinson disease; dementia; muscle diseases that preclude the practice of physical activity; chronic uncontrolled disease (hypertension, diabetes mellitus, chronic pain); unstable cardiovascular disease (acute heart failure, myocardial recent infarction, unstable angina and uncontrolled arrhythmia); using alcohol and other toxic substances; contraindications for performing exercise according the criteria of the American College of Sports Medicine; to practice or have practiced physical exercise program in the last six months; to participate or have participated in regular resistance training (eg, 2-3 times per week) in the previous 12 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Proportion of recurrent fallers (2 or more falls over the study period) | 6 months after completion of the exercise training

SECONDARY OUTCOMES:
Proportion of recurrent fallers (2 or more falls over the study period) | 3 months
Number of falls | 6 months
6-Minute Walk Test (cardiovascular endurance) | 8 weeks
Get Up and Down Test | 8 weeks
10 meters test (gait speed) | 8 weeks
Photometry-measured posture | 8 weeks
Balance Evaluation Systems Test - BESTEST | 8 weeks
Frontal Assessment Battery - FAB | 8 weeks
Quality of life on the Parkinson's Disease Questionnaire-39 - PDQ39 | 8 weeks
World Health Organization Disability Assessment Schedule 2.0 - WHODAS 2.0 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jamary Oliveira-Filho, MD, Principal Investigator — Federal University of Bahia
Locations (1):
- Centro de Referencia Estadual de Atencao a Saude do Idoso (CREASI), Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Duarte GP, Ferraz DD, Trippo KV, Novais MCM, Sales M, Ribeiro NMDS, Oliveira Filho J. Effects of three physical exercise modalities on respiratory function of older adults with Parkinson's disease: A randomized clinical trial. J Bodyw Mov Ther. 2023 Oct;36:425-431. doi: 10.1016/j.jbmt.2023.05.014. Epub 2023 Aug 23. PMID 37949595
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Ferraz DD, Trippo KV, Duarte GP, Neto MG, Bernardes Santos KO, Filho JO. The Effects of Functional Training, Bicycle Exercise, and Exergaming on Walking Capacity of Elderly Patients With Parkinson Disease: A Pilot Randomized Controlled Single-blinded Trial. Arch Phys Med Rehabil. 2018 May;99(5):826-833. doi: 10.1016/j.apmr.2017.12.014. Epub 2018 Jan 11. PMID 29337023